CLINICAL TRIAL: NCT03908333
Title: Phase IB/II Trial of High Dose Ascorbic Acid (AA) + Nanoparticle Paclitaxel Protein Bound + Cisplatin + Gemcitabine (AA NABPLAGEM) in Patients Who Have No Prior Therapy for Their Metastatic Pancreatic Cancer
Brief Title: High Dose Ascorbic Acid and Nanoparticle Paclitaxel Protein Bound and Cisplatin and Gemcitabine (AA NABPLAGEM) in Patients Who Have Metastatic Pancreatic Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Request to close per funding sponsor. Site not moving forward with trial.
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Cancer Research UK (Other); Stand Up To Cancer (Other); Lustgarten Foundation (Other); Destroy Pancreatic Cancer (Other); Translational Genomics Research Institute (Other); HonorHealth Research Institute (Other)
Responsible Party: Principal Investigator, Ben George, Associate Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00034648
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Metastatic Pancreatic Cancer; Pancreatic Cancer; Pancreas Cancer; Pancreatic Adenocarcinoma Resectable; Pancreatic Ductal Adenocarcinoma; Pancreatic Metastasis
Keywords: metastatic pancreatic cancer; cancer; pancreatic; Vitamin C; Ascorbic Acid; Nanoparticle Paclitaxel Protein Bound; cisplatin; gemcitabine; pancreas
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Ascorbic Acid; Taxes; Cisplatin; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Ascorbic Acid Paclitaxel Protein Bound Cisplatin Gemcitabine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AA NABPLAGEM (Experimental): ascorbic acid paclitaxel protein-bound cisplatin gemcitabine
  Interventions: Drug: Ascorbic Acid; Drug: Paclitaxel protein-bound; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Ascorbic Acid — 25, 37.5, 56.25 or 75 grams/m2
  Other Names: Vitamin C
Drug: Paclitaxel protein-bound — 125mg/m2 over 30 minute IV infusions on days 1 and 8 repeated every 21 days
Drug: Cisplatin — 25mg/m2 in 500 mL of NS over 60minute IV infusion on days 1 and 8 repeated every 21 days
Drug: Gemcitabine — 1000mg/m2 in 500 mL over 30 minute IV infusion on days 1 and 8 repeated every 21 days

SUMMARY:
The purpose of this study is to see if a combination of paclitaxel protein bound (also known as nab-paclitaxel), gemcitabine, and cisplatin when given with high dose Ascorbic Acid will be safe and effective in individuals with untreated metastatic pancreatic cancer.

Vitamin C is a nutrient found in food and dietary supplements. It protects cells and also plays a key role in making collagen (which provides strength and structure to skin, bones, tissues and tendons). High-dose vitamin C may be given by intravenous (IV) infusion (through a vein into the bloodstream) or orally (taken by mouth). When taken by intravenous infusion, vitamin C can reach much higher levels in the blood than when the same amount is taken by mouth. Some human studies of high-dose IV vitamin C in patients with cancer have shown improved quality of life, as well as improvements in physical, mental, and emotional functions, symptoms of fatigue, nausea and vomiting, pain, and appetite loss. Intravenous high-dose ascorbic acid has caused very few side effects in clinical trials.

DETAILED DESCRIPTION:
Pancreatic cancer continues to be a very lethal disease. It was estimated that in 2016, 53,070 Americans would be diagnosed with pancreatic ductal adenocarcinoma (PDA), and 41,780 would die from the disease. This makes pancreatic cancer the third leading cause of death from cancer in the US.

PDA is the twelfth most common cancer in the world with 338,000 new cases diagnosed in 2012. It is estimated that worldwide there will be > 300,000 deaths from pancreatic cancer. Furthermore unfortunately PDA is projected to be the second leading cause of death from cancer in the US by 2030.

Detection of pancreatic cancer has notoriously been very late in the disease and therefore the 5-year survival rate is only 8%, which is actually a slight improvement over the last few years. Right now the only potential cure for pancreatic cancer is surgical resection (if the disease is caught early). However only about 20% of PDA patients are eligible for potentially curable resection and unfortunately most (> 80%) have recurrence of their cancer within 2 years of resection, and those recurrences are almost universally fatal.

Recently it has been shown that there are regimens that actually improve survival for patients with advanced stage IV PDA. Conroy and colleagues have developed the Folfirinox regimen, which in a large randomized trial improved survival over gemcitabine as a single agent. Von Hoff and colleagues developed the nanoparticle albumin (nab) associated paclitaxel plus gemcitabine regimen which improved survival over single agent gemcitabine. Even more recently Jameson and colleagues have presented a combined regimen of nab-paclitaxel + gemcitabine + cisplatin in a small 24 patient phase Ib/II trial which showed a response rate of 71% with 2 patients having complete response, a 1-year survival of 65% and a median survival of 16+ months.

While there have been multiple investigators and investigations into the use of ascorbic acid for patients with cancer (see ClinTrials.gov), its use has generally not been found to be of help for patients particularly when given orally - e.g. 10 grams daily.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic pancreatic adenocarcinoma (with measurable disease according to RECIST 1.1 criteria).
* Adequate organ function.
* Have a performance status of 0 or 1 on the ECOG performance scale.
* Female participants of childbearing potential should have a negative serum pregnancy test within 72 hours prior to receiving first dose of study medication.
* Female participants of childbearing potential must be willing to use adequate method of contraception for the duration of the trial through one month after the last dose of trial treatment.
* Male participants must agree to use adequate contraception for the duration of the trial through one month after the last dose of trial treatment.

Exclusion Criteria:

* Patients must have received no previous radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of metastatic disease. Only the following prior treatments in the adjuvant setting are permitted: gemcitabine and/or 5-FU or capecitabine or gemcitabine administered as a radiation sensitizer provided at least six months have elapsed since completion of the last dose and no lingering toxicities are present.
* Palliative surgery less than four weeks prior to initiation of study treatment.
* Exposure to any investigational agent within four weeks prior to initiation of study treatment.
* Patients who need constant use of finger stick blood glucose monitoring for tight control of their diabetes being that the ascorbic acid causes false low readings of glucose via that technology.
* Any person with a G6PD deficiency.
* History of renal oxalate stones (if type of stone is unknown, need to assess urine oxalates level if >60mg/dL, then patient is not eligible for the study).
* Patient is taking acetaminophen at any dose or any medication that contains acetaminophen within 72 hours of first dose of ascorbic acid.
* Hypersensitivity to any of the agents proposed for treatment.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* For female participants: Is pregnant or breastfeeding or expecting to conceive within the projected duration of the trial, starting with the prescreening or screening visit through one month after the last dose of trial treatment.
* For male participants: Is expecting to impregnate a sexual partner within the projected duration of the trial, starting with the prescreening or screening visit through one month after the last dose of trial treatment.
* Patients with evidence of iron overload, defined as a transferrin saturation > 45 percent AND serum ferritin > 200 ng/mL (males) or >150 ng/mL (females).
* Current, serious, clinically significant cardiac arrhythmias as determined by the investigator, or patient receiving a digitalis derivative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 18 weeks
  To determine the maximum tolerated dose (MTD) of high dose ascorbic acid (AA) with triple therapy of nanoparticle paclitaxel protein bound + cisplatin + gemcitabine (NABPLAGEM) in patients with advanced stage IV metastatic pancreatic cancer
Disease Control Rate | 18 weeks
  CR+ PR+SD

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Grade 2-5 Adverse Events assessed using NCI CTCAE v5.0 toxicity criteria | 18 weeks
Progression free survival (PFS) | approximately 12 weeks from last study treatment
  Telephone follow up will be conducted every 12 weeks from the last dose of treatment to determine status of disease progression
Changes in patient's self-reported quality of life: MD Anderson Symptom Inventory (MDASI-GI) | 18 weeks
  Changes in patient's self-reported quality of life will be determined by administering the MD Anderson Symptom Inventory (MDASI-GI)
Changes in patient's self-reported pain levels: Brief Pain Inventory (BPI) | 18 weeks
  Changes in patient's self-reported pain levels will be determined by administering the Brief Pain Inventory (BPI).

CONTACTS AND LOCATIONS:
Overall Officials: Ben George, MD, Principal Investigator — Medical College of Wisconsin
Locations (6):
- United States (6):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - University of California San Diego Moores Cancer Center, San Diego, California
  - Piedmont Cancer Institute, PC, Atlanta, Georgia
  - Piedmont Cancer Institute, PC, Fayetteville, Georgia
  - Piedmont Cancer Institute, PC, Newnan, Georgia
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin